CLINICAL TRIAL: NCT04060901
Title: Compassion-Centered Spiritual Health (CCSH) Interventions for Teams With Faculty and Staff
Brief Title: Compassion-Centered Spiritual Health for Faculty and Staff
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Jennifer Mascaro, Assistant Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IRB00112957
Record Dates: First submitted 2019-08-16; First posted 2019-08-19 (Actual); Last update posted 2020-05-14 (Actual); Status verified 2020-05

CONDITIONS: Health Behavior
Keywords: Spiritual health clinician
MeSH Terms: conditions — Health Behavior

STUDY DESIGN:
Intervention Model Description: CRC teams will be randomized to one of two cohorts; the first cohort will receive the intervention during the first period while the second cohort waits to receive the intervention during the second period.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CCSH Interventions for Teams in Cohort 1 (Experimental): Participants in the first cohort will receive the CCSH Interventions for Teams during the fall session (first intervention period).
  Interventions: Behavioral: CCSH Intervention for Teams
- CCSH Interventions for Teams in Cohort 2 (Experimental): Participants in the second cohort will receive the CCSH Interventions for Teams during the spring session (second intervention period).
  Interventions: Behavioral: CCSH Intervention for Teams

INTERVENTIONS:
Behavioral: CCSH Intervention for Teams — CCSH Interventions for Teams will be a six session intervention. The groups meet once per week for 60 minutes for 4 weeks, coupled with 2 booster sessions over the following 2 months. Participants will receive the CCSH interventional approach, adapted for a group setting, which follows four stages: 1) Preparing the care responder; 2) Attuning to the Relationship; 3) Accessing Compassion, and 4) Entrusting the Careseeker.
  The CCSH approach will be used to assess group dynamics, individual member sources of distress, as well as existing resources for resilience and compassion. Through the intervention, resources will then be identified and accessed in order to respond to team (and individual) sources of distress with greater resilience and increased compassion toward self and others. CCSH clinicians will utilize group process skills to encourage team communication about work-related challenges, enhance team cohesion, and enable interpersonal support among members of the team.

SUMMARY:
Compassion-Centered Spiritual Health (CCSH) at Emory University was launched as a joint creation by Spiritual Health and the Center for Contemplative Science and Compassion-Based Ethics in 2018. The program enhances the practice of spiritual health through CCSH Interventions, which are a Cognitively-Based Compassion Training (CBCT)-based approach to support the practices of spiritual health clinicians. CBCT is a research-based contemplative program developed at Emory University in 2004. CCSH Interventions are provided by spiritual health clinicians across Emory's inpatient and outpatient facilities and beyond, and offer a method to alleviate distress in patients and families and to mitigate burnout in healthcare professionals. While the intervention will be required for some staff and provider populations, Spiritual Health proposes to pilot a voluntary systematic implementation of CCSH Interventions for Teams (CCSH-TI) to clinical research teams at Winship Cancer Institute. Clinical Research Coordinators (CRCs) experience significant emotional and spiritual burden through exposure to patients living with cancer and undergoing clinical trials for cancer treatment. As individuals and teams, CRCs face multiple work-related challenges known to cause distress, including experiences of secondary trauma, exposure to emotional and spiritual suffering of patients and families, and experiences of loss of patients. The researchers of this study hope that offering CCSH Interventions for Teams to CRCs will increase their resilience, wellbeing and compassion toward self and others, with a secondary benefit that burnout will be reduced. By conducting this pilot project, the researchers hope to gain a better understanding of how to optimally implement CCSH for CRC teams at the Winship Cancer Institute.

DETAILED DESCRIPTION:
Previous research indicates that Cognitively-Based Compassion Training (CBCT) improves empathic accuracy, enhances well-being, and attenuates the pro-inflammatory response to psychosocial stress. CBCT is a secularized compassion meditation program adapted from the Tibetan Buddhist mind training (lojong) tradition, and it may be an ideal addendum to the spiritual caregiving provided by Emory University hospital chaplains and chaplain residents to approximately 100,000 patients, staff, and faculty members each year.

With this in mind, The Emory University Spiritual Health department now incorporates CBCT into their training curriculum using a phased approach that began in Fall 2017. The Spiritual Health department also developed an adapted program based on CBCT principles that chaplains can then deliver to patients and staff, called Compassion-Centered Spiritual Health (CCSH). Spiritual Health proposes to pilot a systematic implementation of CCSH Interventions for Teams (CCSH-TI) to clinical research teams at the Winship Cancer Institute.

This is a randomized trial of CCSH Interventions for Teams versus a wait list control condition. CRC teams will be randomized to receive CCSH-TI during a first cohort or to a wait-list group that will receive CCSH-TI during the second cohort. CRCs (n = 93) will be randomized by team to receive CCSH Interventions for Teams either in the fall or in the spring. Participating CRCs will complete self-report measures at 4 timepoints throughout the year: (1) Prior to randomization, (2) immediately upon completion of CCSH Interventions for Teams for cohort 1 (3) prior to CCSH Interventions for Teams for cohort 2, and (4) immediately upon completion of CCSH Interventions for Teams for cohort 2.

ELIGIBILITY:
Inclusion Criteria:

* Emory staff, clinical research coordinators

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2019-08-23 (Actual); Primary Completion 2020-02-07 (Actual); Study Completion 2020-02-07 (Actual)

PRIMARY OUTCOMES:
Change in Professional Quality of Life (ProQOL) Score | Baseline, Week 5, Week 24, Week 29
  The Professional Quality of Life Scale (ProQOL) is a 30-item inventory and is the most commonly used measure of the negative and positive effects of helping others who experience suffering. It has sub-scales for compassion satisfaction, burnout, and compassion fatigue. The sub-scales are summed and converted to t-scores with a mean of 50 and standard deviation of 10. Scores higher than 57 indicate professional satisfaction while scores below 40 indicate possible problems with feeling satisfied professionally.
Staff Retention | Up to Week 29
  Staff retention (number of employees not resigning) will be compared between the teams completing the intervention and those who have not yet participated.
Staff Absenteeism | Up to Week 29
  Staff absenteeism (number of missed work days) will be compared between the teams completing the intervention and those who have not yet participated.

SECONDARY OUTCOMES:
Change in Depression Anxiety and Stress Scale (DASS) Short Form Score | Baseline, Week 5, Week 24, Week 29
  The Depression Anxiety and Stress Scale (DASS) short form is a 21-item likert-scale measure that assesses the frequency of symptoms of depression, anxiety and stress during the past week. Respondents indicate the degree to which they agree with each statement on a scale of 0 to 3 where 0 = does not apply to me at all and 3 = applied to me very much, or most of the time. Total scores range from 0 to 63 and higher scores indicate increased feelings of depression, anxiety and stress.
Change in Revised University of California, Los Angeles (UCLA) Loneliness Scale (R-UCLA) Score | Baseline, Week 5, Week 24, Week 29
  The Revised UCLA Loneliness Scale (R-UCLA) is a 20-item questionnaire measuring general feelings of social isolation and dissatisfaction with one's social interactions. Participants rate each item on a scale from 1 (never) to 4 (often). When scoring the scale, certain items are reversed so that low scores correspond with low loneliness. Total scores range from 20 to 80, where higher scores indicate increased feelings of loneliness.
Change in Patient-Reported Outcomes Measurement Information System (PROMIS) Sleep Disturbance Short Form Score | Baseline, Week 5, Week 24, Week 29
  The PROMIS Sleep Disturbance Short Form is an 8-item scale assessing self-reported perceptions of sleep quality, sleep depth, and restoration associated with sleep. This includes perceived difficulties and concerns with getting to sleep or staying asleep, as well as perceptions of the adequacy of and satisfaction with sleep. Responses are given on a 5-point scale where 1 = no problems and 5 = very problematic. Total raw scores range from 8 to 40 where higher scores indicate greater sleep disturbances.
Change in Connor-Davidson Resilience Scale 25 (CD-RISC-25) Score | Baseline, Week 5, Week 24, Week 29
  The CD-RISC-25 is a 25-item inventory measuring resilience. Responses are on a 5-point scale where 0 = rarely true and 4 = true nearly all of the time. Total scores range from 0 to 100 and higher scores indicate greater resilience.
Change in Nursing Incivility Scale (General, Nurse, and Patient subscales) | Baseline, Week 5, Week 24, Week 29
  The Workplace Incivility Scale is a 43-item instrument assessing perceived disrespect, condescension, or degradation in the healthcare environment. Responses are on a 5-point scale where 1 = strongly disagree and 5 = strongly agree. Total scores for the 3 subscales used here range from 0 to 116 and higher scores indicate greater perceived incivility in the workplace.
Interest in the CCSH Intervention Scale | Baseline or Week 24
  Prior to beginning the CCSH intervention, participants will complete a 6-item questionnaire assessing their interest in learning CBCT. Responses are given on a 7-point scale where 7-point scale where 0 = strongly disagree and 6 = strongly agree. Total scores range from 0 to 36 with higher scores indicating greater interest in the intervention. Participants in Cohort 1 will complete the questionnaire at the Baseline visit and participants in Cohort 2 will complete this questionnaire at the Week 24 visit (prior to beginning the second session of the intervention).
Experiences with the CCSH Intervention Scale | Week 5 or Week 29
  Upon completion of the CCSH intervention the participant's experiences with the intervention will be assessed with a 7-item scale asking questions about how beneficial the intervention was. Responses are given on a 7-point scale where 0 = strongly disagree and 6 = strongly agree. Total scores range from 0 to 42 with higher scores indicating greater satisfaction with the intervention. Participants in Cohort 1 will complete the questionnaire at the Week 5 visit and participants in Cohort 2 will complete this questionnaire at the Week 29 visit.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Mascaro, PhD, Principal Investigator — Emory University
Locations (1):
- Emory University, Winship Cancer Institute, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mascaro JS, Palmer PK, Ash MJ, Peacock C, Sharma A, Escoffery C, Raison C. Feasibility, Acceptability, and Preliminary Effectiveness of a Compassion-Centered Team Intervention to Improve Clinical Research Coordinator Resilience and Well-Being. JCO Oncol Pract. 2021 Jul;17(7):e936-e946. doi: 10.1200/OP.21.00120. Epub 2021 Jun 21. PMID 34152835